CLINICAL TRIAL: NCT03941704
Title: Development of Pre-Packaged Pulse-Based Meals to Ameliorate the Negative Health Consequences of Sedentary Behavior
Brief Title: Pulse-based Foods for Alleviation of Negative Consequences of Sedentary Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 609
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Crossover: 1. Pulse-based diet; 2. Regular diet
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycemic Index (Experimental): Pulse-based diet
  Interventions: Dietary Supplement: Pulse-based diet
- Moderate Glycemic Index (Active Comparator): Regular diet
  Interventions: Dietary Supplement: Regular diet

INTERVENTIONS:
Dietary Supplement: Pulse-based diet — Low Glycemic Index
  Arms: Low Glycemic Index
Dietary Supplement: Regular diet — Moderate Glycemic Index
  Arms: Moderate Glycemic Index

SUMMARY:
The hypothesis is that consumption of pulse-based foods (i.e. containing chickpeas, lentils, and split peas) during the workday will improve insulin sensitivity, glucose tolerance, blood lipids, body composition, and blood pressure in sedentary office workers.One-hundred office workers from a university campus will participate in a cross-over study where they will be randomized (i.e. assigned by chance) to receive pre-packaged pulse-based lunches and snacks to replace their usual lunches/snacks during the work day OR to continue consuming their usual diets for two months. After the first dietary intervention, they will undergo a 1-month "wash-out" and then participate in two months of the opposite dietary intervention. The main outcome to be assessed is change in glucose and insulin (i.e. blood sugar control) determined during an oral glucose tolerance test. Secondary outcomes include changes in body composition, lipids, and blood pressure.

During the pulse-based diet phases, participants will be supplied with a ready-to-eat lunch and two snacks to eat during each workday. These will contain a total of 150g/d dry weight (250g/d wet weight) pulses

DETAILED DESCRIPTION:
Sedentary behaviour has been deemed the "new smoking" based on multiple and potent negative impacts on health. Moreover, sedentary behaviour is a strong predictor of type 2 diabetes risk and cardiovascular disease. Previous studies have show that pulse-based meals derived from lentils, beans, chickpeas, and peas are effective for alleviating risk factors associated with diabetes and cardiovascular disease in clinical populations including older adults, overweight and obese individuals, and women with polycystic ovary syndrome; however, to date, there have been no nutrition-based interventions for alleviating risk factors for diabetes specifically targeting office workers exposed to long periods of sitting. Although people are aware of the health benefits of pulses, a major barrier to increased consumption continues to be a lack of knowledge on how to prepare pulse-based meals. This proposed study is designed to overcome this barrier. The main goal of this research study is to determine whether improvements in cardio-metabolic health can be realized by giving people pulse-based lunches and snacks to replace their regular workplace lunches and snacks. In this randomized controlled trial, 100 office workers from the University of Saskatchewan will participate in a cross-over study where they will be randomized into one of two diets for 2 months: Receive pre-packaged pulse-based lunches and snacks to replace their usual lunches/snacks during the work day OR to continue consuming their usual diets for two months. After a one-month washout, they will cross-over to the other condition. The primary outcome measure, Matsuda Index (determined by blood glucose and insulin responses to an oral glucose tolerance test), will be assessed before each diet phase and at the end (i.e. two months) of each diet phase. Secondary outcome measures (body composition, waist girth, lipids, blood pressure will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* 18y or older
* Engaged in >5 hours per day sitting

Exclusion Criteria:

* Diagnosed with diabetes
* taking glucose or lipid-lowering medication
* Regular consumers of pulses (1.5 cups (250g) or greater of pulses per week)
* Engaged in 60 minutes or greater of physical activity per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from baseline to 8 weeks
  Matsuda Index determined by glucose and insulin response to oral glucose tolerance test

SECONDARY OUTCOMES:
Glucose area under the curve | Change from baseline to 8 weeks
  Glucose area under the curve from a 2-hour oral glucose tolerance test
Insulin area under the curve | Change from baseline to 8 weeks
  Insulin area under the curve from a 2-hour oral glucose tolerance test
Fasting glucose | Change from baseline to 8 weeks
  Fasting glucose
Fasting insulin | Change from baseline to 8 weeks
  Fasting insulin
Low-density lipoprotein cholesterol | Change from baseline to 8 weeks
  LDL-C from fasting blood samples
High-density lipoprotein cholesterol | Change from baseline to 8 weeks
  HDL-C from fasting blood samples
Total cholesterol | Change from baseline to 8 weeks.
  Total cholesterol from fasting blood samples
Triglycerides | Change from baseline to 8 weeks
  Triglycerides from fasting blood samples
Waist Girth | Change from baseline to 8 weeks
  Waist Girth
Fat mass | Change from baseline to 8 weeks
  Fat mass from DXA measurements
Lean tissue mass | Change from baseline to 8 weeks
  Lean tissue mass from DXA measurements
Systolic blood pressure | Change from baseline to 8 weeks
  Systolic blood pressure measured at rest
Diastolic blood pressure | Change from baseline to 8 weeks
  Diastolic blood pressure measured at rest

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No